CLINICAL TRIAL: NCT03169920
Title: Evaluation of the Efficacy of Autologous Platelet Rich Fibrin With Modified Minimally Invasive Surgical Technique (M-MIST) in the Treatment of Intrabony Defects: A Randomized Clinical Trial
Brief Title: Efficacy of PRF With M-MIST in the Treatment of Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nabeela perio
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Modified-Minimally Invasive Surgical Technique + PRF
  Interventions: Procedure: Modified-Minimally Invasive Surgical Technique + PRF
- Control Group (Active Comparator): Modified-Minimally Invasive Surgical Technique alone.
  Interventions: Procedure: Modified-Minimally Invasive Surgical Technique

INTERVENTIONS:
Procedure: Modified-Minimally Invasive Surgical Technique + PRF
  Arms: Test Group
Procedure: Modified-Minimally Invasive Surgical Technique
  Arms: Control Group

SUMMARY:
This study evaluates the efficacy of M-MIST with or without PRF in the treatment of intrabony defects.Taking into consideration of advantages of PRF and M-MIST it was hypothesised that this combination (PRF+M-MIST) would be more beneficial in achieving healing of intrabony defects. Furthermore the concomitant use of Platelet Rich Fibrin with M-MIST has not been previously attempted in periodontal practice.

DETAILED DESCRIPTION:
INTRODUCTION

In the last two decades, some clinical investigators have focused their interest on the development of minimally invasive surgical approaches in periodontal surgery. Harrel & Rees proposed the minimally invasive surgery (MIS) with the aim to produce minimal wounds, minimal flap reflection and gentle hand ling of the soft and hard tissues in periodontal surgery. Cortellini & Tonetti tested the use of operative microscopes and microsurgical instruments to increase visual acuity and accuracy in the application of papilla preservation flaps in periodontal regeneration. The increased patient acceptance and decreased morbidity with minimally invasive surgery offers a promising therapeutic modality and may replace the need for more extensive surgical procedures. Recently, a new surgical approach, the ''minimally invasive surgical technique (MIST)'', has been proposed to treat isolated intrabony defects with periodontal regeneration. Results from a cohort study in isolated deep intrabony defects showed marked improvements in terms of clinical attachment level (CAL) gains and PD reduction. The background foundations for this technique are the concepts of the MIS, and the application of papilla preservation techniques with a microsurgical approach. The cited study also reported a very limited patient morbidity and a reduced length of the surgical procedure following application of the MIST. An enhancement of this technique, the modified minimally invasive surgical technique (M-MIST), has been recently designed to further reduce the surgical invasiveness, with three major objectives in mind: (1) minimize the interdental tissue tendency to collapse, (2) enhance the wound/soft tissue stability and (3) reduce patient morbidity.

Periodontal researchers and clinicians, in an effort to develop effective regenerative therapies, have sought to understand key events involved in the regeneration of the periodontium. An increased knowledge of specific cellular response and function within the periodontium has led to the development of numerous treatment modalities exhibiting different degrees of success.

Treatments including ''grafting'' with bone or bone substitutes, stimulation of cells with growth factors, hormones, or extracellular matrix proteins; cell occlusive barrier membranes for selective cell growth in periodontal defects; and modification of the tooth root surface have all been explored for their ability to predictably regenerate the periodontium. Although some treatments have yielded promising results, there remains a need for a treatment that leads to faster and more predictable regeneration of the periodontium.

The development of bioactive surgical additives, which are being used to regulate the inflammation and increase the speed of healing process, is one of the great challenges in clinical research. In this sense, healing is a complex process, which involves cellular organization, chemical signals, and the extracellular matrix for tissue repair. The understanding of healing process is still incomplete, but it is well known that platelets play an important role in both hemostasis and wound healing processes.

Platelets' regenerative potential was introduced in the 70's, when it was observed that they contain growth factors that are responsible for increase collagen production, cell mitosis, blood vessels growth, recruitment of other cells that migrate to the site of injury, and cell differentiation induction, among others.

One of the latest innovations in oral surgery is the use of platelet concentrates for in vivo tissue engineering applications. Platelet concentrates are a concentrated suspension of growth factors found in platelets, which act as bioactive Platelet rich fibrin (PRF) was first used in 2001 by Choukroun et al., specifically in oral and maxillofacial surgery, and is currently considered as a new generation of platelet concentrate. It consists of a matrix of autologous fibrin and has several advantages over Platelet rich plasma (PRP), including easier preparation and not requiring chemical manipulation of the blood, which makes it strictly an autologous preparation.

PRF consists of an autologous leukocyte-platelet-rich fibrin matrix, composed of a tetra molecular structure, with cytokines, platelets, cytokines, and stem cells within it, which acts as a biodegradable scaffold that favors the development of microvascularization and is able to guide epithelial cell migration to its surface. Also, PRF may serve as a vehicle in carrying cells involved in tissue regeneration and seems to have a sustained release of growth factors in a period between 1 and 4 weeks, stimulating the environment for wound healing in a significant amount of time. It has a complex architecture of strong fibrin matrix with favorable mechanical properties and is slowly remodeled, similar to blood clot . Some studies have demonstrated that PRF is a healing biomaterial with a great potential for bone and soft tissue regeneration, without inflammatory reactions and may be used alone or in combination with bone grafts, promoting hemostasis, bone growth, and maturation. This autologous matrix demonstrated in in vitro studies a great potential to increase cell attachment and a stimulation to proliferate and differentiate osteoblasts. Dohan et al. stated that PRF has immunological and antibacterial properties, may lead to leukocyte degranulation, and has some cytokines that may induce angiogenesis and pro/anti-inflammatory reactions.

Taking into consideration of above mentioned advantages of PRF and M-MIST it was hypothesised that this combination (PRF+M-MIST) would be more beneficial in achieving healing of intrabony defects. Furthermore the concomitant use of Platelet Rich Fibrin with M-MIST has not been previously attempted in periodontal practice. Thus the aim of the study is to evaluate the efficacy of PRF along with M-MIST in the treatment of intrabony defects.

MATERIAL AND METHOD

This study will be conducted in Department of Periodontics and Oral Implantology , Post Graduate Institute Of Dental Sciences,(PGIDS) Rohtak, Haryana.

STUDY POPULATION

Patients will be recruited from regular outpatient department of the Department of Periodontics and Oral Implantology. Minimum total 36 patients will be included as per eligibility in this study.

Prior informed consent will be taken from each patient after explaining the procedure in patient's language along with risk and benefits involved.

METHODOLOGY

Sample size and randomization

A total number of 36 patients were selected and divided into 2 groups of 18 each

All the eligible patients will be randomly assigned at the time of surgery into either of the two groups:

* Test group: Modified-Minimally Invasive Surgical Technique + Platelet Rich Fibrin
* Control group: Modified-Minimally Invasive Surgical Technique alone.

Clinical parameters

All the clinical parameters will be recorded at baseline, 3 months and 6 months post-surgery.

Gingival status will be assessed using the Loe and Silness Gingival Index . Plaque status will be recorded using Silness and Loe Plaque Index. The clinical parameters will include relative clinical attachment level (CAL), probing pocket depth (PPD) and gingival recession will be recorded to the nearest millimetre (at the deepest location of the selected interproximal site) with the help of a UNC-15 probe (university of north carolina)at baseline, 3 months and 6 months post-surgery.

All the parameters will be clinically assessed by a single examiner.

Radiographic parameters

Intra-oral periapical radiographs of the selected teeth will be taken using long cone paralleling technique at baseline, 3 months and 6 months post-surgery.

All the radiographs will be assessed by the another investigator.

The anatomical landmarks of the intrabony defect will be selected on the radiographs based on the criteria set by Schei et al., which include cementoenamel junction (CEJ), alveolar crest (AC) and base of the defect (BD). The radiographic parameters evaluated will be percentage bone fill (%BF) and the change in alveolar crest position (C-ACP).

Surgical approach (M-MIST)

All the surgical procedures will be performed using microsurgical instruments. The defect-associated papilla will be surgically approached with the M-MIST . The defect associated papilla will be surgically approached with modified papilla preservation technique at interdental sites. A thorough surgical debridement of the osseous defect will be performed using curettes from under the papilla, aided with surgical microscope. The defect will be debrided with mini curettes and the root will be carefully planed. Special care will be taken to reach all the parts of the exposed root surface and residual bony wall partly hidden by the non elevated lingual and papillary soft tissue. To allow instrumentation the buccal papillary flap will be slightly reflected carefully protected with a periosteal elevator and frequently irrigated with saline. Once the debridement is over, the vertical defect depth (from the bottom of the defect to the alveolar crest) and the number of bony walls present will be recorded. If the vertical defect depth is ≥3 mm, final subject eligibility will be confirmed. The required quantity of the PRF will be delivered into the osseous defect in test group.

Post-surgical care

Appropriate post-operative instructions will be given to the patients. Sutures will be removed 1 week following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy chronic periodontitis patients
* Presence of one tooth with probing depth (PD) and clinical attachment loss (CAL) ≥5 mm associated with an interdental intrabony defect depth of≥3 mm.
* Only patients with optimal compliance, as assessed during the cause-related phase of therapy, will be selected.
* Cause related therapy (CRT) including scaling and root planning will be performed and oral hygiene instructions will be given to all the study subjects.

Exclusion Criteria:

* Systemic illness (chronic inflammatory diseases like diabetes mellitus, arthritis, history of viral infection or pyrexia over the past one month) known to affect the periodontium or outcome of periodontal therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Patients having history of receiving antibiotics or periodontal treatment over the past 3 months.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Pregnant or lactating mothers.
* Smokers and tobacco chewers.
* Fractured/perforated roots.
* Teeth with mobility greater than grade II (Miller 1943) and furcation involvement (class II and class III, Glickman 1953) or with clinical signs of untreated acute infection at surgical site, apical pathology, and severe root irregularities will be excluded.

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
PD | 6 months
  pocket depth
CAL | 6 months
  clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Nabeela Ahmed, Principal Investigator — Post Graduate Institute of Dental Sciences, Rohtak. HARYANA .INDIA; SHIKHA TEWARI, Study Chair — Post Graduate Institute of Dental Sciences, Rohtak. HARYANA .INDIA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmad N, Tewari S, Narula SC, Sharma RK, Tanwar N. Platelet-rich fibrin along with a modified minimally invasive surgical technique for the treatment of intrabony defects: a randomized clinical trial. J Periodontal Implant Sci. 2019 Oct 9;49(6):355-365. doi: 10.5051/jpis.2019.49.6.355. eCollection 2019 Dec. PMID 31886028